CLINICAL TRIAL: NCT06240468
Title: Dynamic Changes in Human Microbiome Predict the Risk of Adverse Outcomes in Patients With Acute Ischemic Stroke: a Multicenter Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CALM2003
Record Dates: First submitted 2023-08-11; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-05

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, stool, mouth swab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AIS patient: AIS inclusion criteria
  (1) Inclusion criteria
  1. Meet the diagnostic criteria for AIS or TIA;
  2. Age 18-80 years old;
  3. within 7 days of the onset of stroke;
  4. Sign informed consent, provide relevant medical history and biological specimens;
  5. Have lived in the local city for the last three years.
  (2) Exclusion criteria
  1. Patients with recurrent stroke within the past year when first enrolled;
  2. mRS > 2 points before stroke onset;
  3. malignant tumor;
  4. Liver and kidney dysfunction (alanine aminotransferase or aspartate aminotransferase >2 times the upper limit of normal, creatinine > 1.5 times the upper limit of normal);
  5. History of drug abuse and chemical poisoning (e.g. pesticide poisoning);
  6. In the acute stage of stroke (within 7 days from the onset of stroke) stool specimens could not be collected.
  Interventions: Other: not have
- Cognitive/emotional subcohort: (I) Inclusion criteria:
  1. It has been included in the AIS queue, meeting the inclusion criteria of the main AIS queue;
  2. NIHSS≤15; (II) Exclusion criteria:
  (1) Patients with aphasia and unable to cooperate in completing the cognitive/emotional assessment during the study; (2) previous severe mental disorder and dementia (AD8 scale score ≥2); (3) A history of severe anxiety and depression; (4) Previous history of seizures.
  Interventions: Other: not have
- healthy person: health
  Interventions: Other: not have

INTERVENTIONS:
Other: not have — not have

SUMMARY:
(1) The main purpose

To explore the predictive value of human microbiome and its metabolome for adverse prognosis in patients with acute ischemic stroke (AIS).

(2) Secondary purposes

1. To explore the characteristics of cross-regional disturbance of human microbiome in stroke patients;
2. To investigate the characteristics and rules of bacterial flora changes before and after recurrent apoplexy;
3. Markers closely related to AIS prognosis and cognitive emotional complications were excavated by metagenomic, metabolic, peptide and imaging groups.
4. To explore the relationship between serum markers of ultra early stage and prognosis.

DETAILED DESCRIPTION:
This is a multicenter, prospective clinical cohort study. In this study, 2000 patients with AIS were continuously enrolled in a multicenter study, and neurological function scores (including NIHSS, mRS And ADL scores) were evaluated during and after hospitalization (3 months, 6 months, 12 months) by outpatient/telephone follow-up, and recurrent stroke and other cardiovascular and cerebrovascular events were recorded. Besides, periodontal swabs, urine, feces and blood samples were collected at multiple time points (Residual blood after the first clinical examination was collected for patients with very early stage, and blood, urine, feces and periodontal swabs were collected the next day after admission, before discharge, 3 months and 6 months after admission. Since the collection time of fecal specimens is difficult to control, only two specimens should be collected 48 hours apart during hospitalization. The first specimen should be collected as early as possible, and the time of specimen separation should be recorded.

Baseline data collection and discharge neurological function score were completed for the enrolled AIS patients before discharge, and the final diagnosis, stroke etiology classification, lifestyle survey (1 year ago), and relevant examination and treatment during hospitalization were recorded. Neurological function score, lifestyle survey, new cardiovascular and cerebrovascular events and biological specimen collection (blood, urine, feces, periodontal swab) were recorded during outpatient visits 3 months and 6 months after admission. Telephone follow-up was conducted 12 months after admission, mRS Score, ADL score and new cardiovascular and cerebrovascular events were recorded.

For the patients (750 cases) who met the criteria for inclusion in the cognitive emotion subcohort, outpatient emotional and cognitive psychological assessment was also required before discharge, 3 months and 6 months after admission on the basis of the AIS cohort.

For the subcohort with recurrence within 1 year, only data collection during hospitalization (baseline hospitalization data) and biological specimen collection during hospitalization (residual blood after the first laboratory examination was retained for patients in the very early stage, and blood, urine, feces, and periodontal swabs were collected the next day after admission and before discharge. As the time of fecal sample collection is difficult to control, it only needs to be 48 hours between hospitalization), and no follow-up will be conducted after discharge.

In addition, 500 patients without stroke were recruited as healthy control group according to the prescribed inclusion criteria.

No randomization or any study protocol-driven treatment will be administered or provided to the subject during the study. If clinically applicable, treatment decisions and treatment options are made at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for AIS or TIA
* Age 18-80 years old
* Within 7 days of the onset of stroke
* Sign informed consent, provide relevant medical history and biological specimens
* Have lived in the local city for the last three years

Exclusion Criteria:

* Patients with recurrent stroke within the past year when first enrolled
* mRS > 2 points before stroke onset
* malignant tumor
* Liver and kidney dysfunction (alanine aminotransferase or aspartate aminotransferase >2 times the upper limit of normal, creatinine > 1.5 times the upper limit of normal)
* History of drug abuse and chemical poisoning (e.g. pesticide poisoning)
* In the acute stage of stroke (within 7 days from the onset of stroke) stool specimens could not be collected

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
All scale surveys were completed at 3, 6 and 12 months after admission | The evaluation time was during admission, three months follow-up, six months follow-up and twelve months follow-up.
  To evaluate the prognosis of neurological function (mRS, NIHSS), the incidence of new cardiovascular and cerebrovascular events and death (any stroke /TIA/ myocardial infarction) at admission and 3, 6 and 12 months after admission;To evaluate the prognosis of neurological function (mRS, NIHSS), the incidence of new cardiovascular and cerebrovascular events and death (any stroke /TIA/ myocardial infarction) at admission and 3, 6 and 12 months after admission;
Number of participants with recurrent stroke within one year of follow-up period | The follow-up period is one year.
  Participants who had recurrent stroke and were readmitted within one year of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China